## TRANSCENDENCE RESEARCH: Holistic Education For Colonized Countries Primarily English Speaking

NCT06098755

October 2, 2025

## **SEXUAL CONSENT FORM**

| I. THE PARTIES. This Sexual Cons, 20 | sent Form ("Consent Agreement") is made<br>between: |
|---|---|
| Proposer: | ("Proposer") |
| AND | |
| Consenter: | ("Consenter"). |
| | Consenter are sexually attracted to each other and ttraction through participation in one or more sexual |
| each other for the aforesaid purpose, 20 | and the Proposer make their bodies available to e from time: □ AM □ PM on the date of (today's date if left blank) for a period of |
| hours, during which period they con | sent to participate in the following activities. |
| III. ACTIVITIES. (initial all that apply | <b>/</b> ) |
| Proposer / Consenter | |
| / Digital penetrat / Digital penetrat / Digital penetrat / Oral sex (received) / Oral sex (giving) / Vaginal sex (received) / Anal sex (received) / Anal sex (giving) / Restraint, using | without the insertion of tongue into mouth ion (receiving in (specify orifice(s))) ion (giving in (specify orifice(s))) ving) g) ceiving: females only) ving) g: males only or females with toys) g the following devices (specify) g devices in or on the body (specify) |
| IV. CONTRACEPTION. | |
| The <b>Proposer</b> is using the following | g methods of contraception on an ongoing basis: |
| The <b>Proposer</b> will use the following vaginal/anal* penetrative activities: | methods of contraception and/or protection during |
| The Consenter is using the following | ng methods of contraception on an ongoing basis: |
| The <b>Consenter</b> will use the followin vaginal/anal* penetrative activities: | ng methods of contraception and/or protection during |



| | age in activities heretofore | oon sexual activities, and that both parties not consented to, the parties agree as |
|---|---|---|
| | s Consent Agreement with | y kind other than that specified and hout the establishment of a new, separate |
| Initiale | ed (Proposer) | Initialed (Consenter) |
| Form shall be pres | umed to be <b>consented to</b> | specified and consented to in this Consent of with the retroactive checking of the gning of this Consent Form. (See clause 1 |
| Initiale | ed (Proposer) | Initialed (Consenter) |
| Form shall be pres | umed to be consented to | specified and consented to in this Consent<br>by <b>mutual verbal consent</b> during the<br>n in the present Consent Form. (See |
| Initiale | ed (Proposer) | Initialed (Consenter) |

V. RATCHET CLAUSE. Whereas the Proposer and the Consenter are aware that

Clause 1. Whereas both Proposer and Consenter recognize that alternatives a) and b) are likely significantly to disrupt any activities consented to under this Consent Agreement;

Therefore, the Proposer and the Consenter further agree that should the disruption of agreed activities, caused by the making of a further Consent Agreement (under a) above) or the retroactive amendment of this Consent Agreement (under b) above), result in a loss of desire to continue the activities herein consented to, consent for those activities consented to herein may/may not\* be withdrawn by the verbal statement of one of the parties to this Consent Agreement.

Clause 2. Whereas both Proposer and Consenter recognize that alternative c) involves verbal consent of which no physical evidence will exist thereafter; Therefore, the Proposer and the Consenter further agree that such consent shall/shall not\* be recorded using an audio recording device; and Whereas both Proposer and Consenter recognize that should no audio recording of verbal consent under this ratchet clause be made, neither party could subsequently prove affirmative consent to the activities that were verbally agreed upon; Therefore, both parties hereby waive their right to claim that no such affirmative consent was given. Equivalently, the Proposer and the Consenter hereby consent to any further activities that can be reasonably deemed to follow naturally from the activities herein consented to.